CLINICAL TRIAL: NCT03309982
Title: A Randomized Placebo-controlled Cross-over Design Study Investigating the Effects of a Plant Polyphenol Blend on the Intestinal Inflammatory and Metabolic Responses to a High Fat Meal in Healthy Subjects
Brief Title: Intestinal Inflammatory and Metabolic Responses to a High Fat Meal and Plant Polyphenol Blend
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Responsible Party: Principal Investigator, Patricia Oteiza, PhD, Professor, University of California, Davis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 17-PHX-0002
Record Dates: First submitted 2017-10-04; First posted 2017-10-16 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Anthocyanins

STUDY DESIGN:
Intervention Model Description: A randomized placebo-controlled cross-over design study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant polyphenol blend (Experimental): The study product (4 g) consists of 3 g of a mix a maltodextrins, and 1 g of anthocyanin-rich plant polyphenol blend containing: 1) 100 mg bilberry extract; 2) 300 mg black currant extract; and 3) 600 mg black rice extract.
  Interventions: Dietary Supplement: Plant polyphenol blend
- Placebo (Placebo Comparator): The placebo (4 g) consists of a mix of maltodextrins (3.85 g) and Red Dye No. 40 (0.125 g) and Blue Dye No. 1 (0.025 g).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Plant polyphenol blend — A powder product that will be mixed into a drink and consumed immediately prior to eating a high-fat meal
  Arms: Plant polyphenol blend
Other: Placebo — A powder product that will be mixed into a drink and consumed immediately prior to eating a high-fat meal
  Arms: Placebo

SUMMARY:
This study will investigate the beneficial effects of supplementation with a plant polyphenol blend rich in anthocyanins on parameters of inflammation and metabolic responses following a challenge with a high-fat (HF) meal.

The investigators will use a randomized crossover study to investigate the effects of: 1) placebo (control); 2) plant polyphenol blend rich in anthocyanins; on systemic inflammatory markers (endotoxemia, cytokines, NF-κB), glucose and lipid metabolic responses following consumption of a high-fat (HF) meal in healthy subjects. The high-fat meal (320 g) consists of English muffin bread, sausage, egg and cheese, obtained from US market and completed with palm fat. The total energy content of the high-fat meal is 1,026 Kcal with 70.5 g of fat (29.8 g of saturated fat), 270 mg of cholesterol, 65 g carbohydrate, 5.2 g sugar, and 33 g protein with a total of 62% energy originated from fat, 25% from carbohydrates and 13% from protein. The high-fat meal will be standard and it will not be adjusted for large and small participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects who, in the opinion of the investigator, are free of any medical conditions that might affect study measures.
2. Males and females
3. Age between 18 - 35 years inclusive
4. Subjects with BMI of 22 - 29.9 kg/m2
5. Subjects who agree to discontinue the use of pre- and probiotic and/or polyphenol supplements from 4 weeks prior to the first and through the last study visit
6. Subjects who agree to discontinue foods containing anthocyanins (such as blueberries, blackberries, bilberries, cherries, grapes, grape juice, pomegranate, raspberries, huckleberries, strawberries, and red wine) for at least 1 week prior to each visit.
7. Subjects with no known allergies to study product or components (bilberries, black currants, rice)
8. Subjects willing to completely consume high-fat meal and assigned study product
9. Subjects willing to consume a similar, low fat/low flavonoid \dinner the evening before each high-fat meal visit
10. Subjects have given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Age < 18 or > 35 years
2. BMI < 22 or > 29.9 kg/m2
3. Vegetarian or other dietary restrictions that would not allow the subject to consume the highfat meal
4. Regularly participates in endurance exercise activities (e.g. marathon running, triathlons)
5. Uncontrolled hypertension defined as diastolic blood pressure ≥ 95 mmHg or systolic blood pressure ≥ 160 mmHg
6. Screening serum triglycerides > 150 mg/dL
7. Screening fasting blood glucose < 50 mg/dL or > 100 mg/dL
8. Current smoker or use of tobacco products within the past year
9. Individuals who binge drink (alcohol intake ≥ 5 alcoholic drinks for males or ≥4 alcoholic drinks for females on the same occasion (i.e., at the same time or within a couple of hours of each other)
10. Substance abuse or dependence within the prior 60 days.
11. Daily use of anti-inflammatory medications including NSAIDs and aspirin in the last 4 weeks
12. Use of laxative medications or other products that promote colon cleansing in the last 4 weeks
13. History of restricted diets or use of herbal supplements or medications that interfere with insulin metabolism in the last 4 weeks
14. History of stroke, hepatic, kidney, thyroid disease or cancer
15. History of immune related disorders or Raynaud's disease
16. Current clinically significant depression, anxiety or other psychiatric condition
17. History of malabsorption or GI tract disorders
18. History of GI surgeries (i.e. lapband, gastric bypass, etc.)
19. Diarrhea or oral antibiotic intake within the last 4 weeks
20. Weight change (> 5%) in the last 8 weeks
21. Subject with known history of eating disorders such as bulimia, anorexia, or muscle dysmorphia
22. Allergy or sensitivity to the study product or components of the high-fat meal
23. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma endotoxin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure endotoxin in plasma

SECONDARY OUTCOMES:
Change from baseline in plasma IL-6 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure IL-6 in plasma
Change from baseline in plasma insulin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure insulin in plasma
Change from baseline in plasma GLP-1 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure GLP-1 in plasma
Change from baseline in plasma GLP-2 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure GLP-2 in plasma
Change from baseline in plasma GIP at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure GIP in plasma
Change from baseline in plasma adiponectin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure adiponectin in plasma
Change from baseline in plasma leptin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure leptin in plasma
Change from baseline in plasma ghrelin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure ghrelin in plasma
Change from baseline in plasma triglycerides at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure triglycerides in plasma
Change from baseline in plasma total cholesterol at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure total cholesterol in plasma
Change from baseline in plasma HDL at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure HDL in plasma
Change from baseline in plasma LDL at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure LDL in plasma
Change from baseline in plasma zonulin at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure zonulin in plasma
Change from baseline in plasma total polyphenols at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure total polyphenols in plasma
Change from baseline in plasma total anthocyanidins at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure total anthycyanidins in plasma
Change from baseline in plasma total catechins at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure total catechins in plasma
Change from baseline in plasma glucose at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure glucose in plasma
Change from baseline in PBMC IL-8 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure IL-8 in PBMC
Change from baseline in PBMC IL-10 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure IL-10 in PBMC
Change from baseline in PBMC IL-1β at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure IL-1β in PBMC
Change from baseline in PBMC IL-12p70 at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure IL-12p70 in PBMC
Change from baseline in PBMC TNFa at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure TNFa in PBMC
Change from baseline in PBMC NF-kB at 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption | Baseline, 0.5 hr, 1 hr, 2hrs, 3hrs, and 5hrs post high-fat meal consumption
  blood sample collected by venipuncture to measure NF-kB in PBMC
Change from baseline in fingerstick triglycerides at 15 minutes post high-fat meal consumption | Baseline, and 15 minutes post high-fat meal consumption
  blood sample collected by fingerstick to measure triglycerides
Change from baseline in fingerstick total cholesterol at 15 minutes post high-fat meal consumption | Baseline, and 15 minutes post high-fat meal consumption
  blood sample collected by fingerstick to measure total cholesterol
Change from baseline in fingerstick HDL at 15 minutes post high-fat meal consumption | Baseline, and 15 minutes post high-fat meal consumption
  blood sample collected by fingerstick to measure HDL
Change from baseline in fingerstick LDL at 15 minutes post high-fat meal consumption | Baseline, and 15 minutes post high-fat meal consumption
  blood sample collected by fingerstick to measure LDL
Change from baseline in fingerstick glucose at 15 minutes post high-fat meal consumption | Baseline, and 15 minutes post high-fat meal consumption
  blood sample collected by fingerstick to measure glucose

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Oteiza, PhD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Nutrition Department, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No